CLINICAL TRIAL: NCT06106282
Title: Breast Cancer Survivors Who Experience Aromatase Inhibitor Associated Musculoskeletal Symptoms (AIMSS): A Multidisciplinary Pain Program Designed to Decrease Pain and Improve Functioning, Mood, and Medication Adherence.
Brief Title: Breast Cancer Survivors Who Experience Aromatase Inhibitor Associated Musculoskeletal Symptoms (AIMSS)
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 23-003085; NCI-2023-06241 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-003085 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Hormone Receptor-Positive Breast Carcinoma
MeSH Terms: conditions — Breast Carcinoma In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients attend a 2-day treatment program and complete questionnaires on study. Patients also have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study evaluates the effectiveness of a cognitive behavioral multicomponent treatment program in improving pain, mood, and functioning while reducing medication non-adherence in breast cancer patients with Aromatase Inhibitor Associated Musculoskeletal Symptoms (AIMSS).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the effectiveness of a Multidisciplinary Pain Program for AIMSS, specifically determine the impact of the program on level of pain, functional status, and adherence to prescribed medication.

II. To identify predictors of improvement in pain, functional status, and mood following participation in the program.

OUTLINE: This is an observational study.

Patients attend a 2-day treatment program and complete questionnaires on study. Patients also have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients are 18 years old or more.

  * A breast cancer survivor ECOG =< 2, stage 0-III HR+ who is experiencing musculoskeletal symptoms associated with aromatase inhibitors intake
  * Patients must be at least 6 months on aromatase inhibitors and for no more than 7 years

Exclusion Criteria:

* Breast cancer survivor patients that are not in aromatase inhibitor treatment or have less than 6 months of treatment or more than 7 years of treatment.

  * Asymptomatic patients
  * Patients less than 18 years old
  * Patient that are not being followed as a Mayo Clinic patient

    * Patients with stage IV breast carcinoma
    * Patients that are HR -
    * Patients that are ECOG 3 or more

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage 0-III HR+ breast cancer and AIMSS (Aromatase Inhibitor Associated Musculoskeletal Symptoms) at Mayo Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Adherence to Aromatase Inhibitor (AI) treatment regimen | Baseline; up to 12 months post-treatment
  Adherence to AI treatment regimen will be recorded based on self-report. Patient self-report will categorize each subject as adherent or non-adherent to AI medication. Baseline and follow-up data from each timepoint will be compared to evaluate treatment impact on outcomes.
Functional impairment (quality of life) | Baseline; up to 12 months post-treatment
  Functional impairment (quality of life) will be assessed using the Symptom Impact Questionnaire (SIQR), which has three domains: Function, Overall and Symptoms. Domain 1 (Function) consists of 9 questions answered on a scale where respondent choose a box between "No difficulty" and "Very difficult." Domain 2 (Overall) consists of 2 questions answered on a scale where respondent choose a box between "Never" and "Always." Domain 3 (Symptoms) consists of 10 questions answered on a scale where respondents choose a box between two extremes (e.g., No pain/Unbearable pain or Awoke rested/Awoke very tired). Baseline and follow-up data from each timepoint will be compared to evaluate treatment impact on outcomes.
Fatigue | Baseline; up to 12 months post-treatment
  Fatigue will be measured using the Brief Fatigue Inventory (BFI) from MD Anderson. The BFI is a nine-question scale in which respondents rate each item on a 0-10 numeric scale, with 0 meaning "no fatigue" and 10 meaning "fatigue as bad as you can imagine." Baseline and follow-up data from each timepoint will be compared to evaluate treatment impact on outcomes.
Level of pain | Baseline; up to 12 months post-treatment
  Level of pain will be assesses using the Pain Catastrophizing Scale (PCS). The PCS is a 13-item self-report questionnaire answered using a 5-point Likert scale ranging from 0 (never) to 4 (always). The final score is categorized as rumination, magnification, or helplessness.Baseline and follow-up data from each timepoint will be compared to evaluate treatment impact on outcomes.
Mood | Baseline; up to 12 months post-treatment
  Mood/depression will be assessed using the Center for Epidemiologic Studies Depression Scale Revised (CES-D-R). The CES-D-R is a 20-question survey with 4 available answers for each question: Rarely or none of the time (less than 1 day); Some or a little of the time (1-2 days); Occasionally or a moderate amount of time (3-4 days); or Most or all of the time (5-7 days). Baseline and follow-up data from each timepoint will be compared to evaluate treatment impact on outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara K. Bruce, Ph.D., L.P., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials